CLINICAL TRIAL: NCT07223099
Title: Sauna for Offline Connections and Interactive, Authentic Living
Acronym: SOCIAL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Tiny Blue Dot Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SOCIAL
Record Dates: First submitted 2025-10-29; First posted 2025-10-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Loneliness
Keywords: Loneliness; Sauna; Gen Z; Young adult; Emerging adult

STUDY DESIGN:
Intervention Model Description: All participants will receive the weekly sauna visit intervention (2-hour visits to a sauna in San Francisco, either alone or with one person of their choice) for 8 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sauna Visits (Experimental): Participants will complete 2-hour visits, by themselves or with another person of their choosing, to a local sauna in San Francisco for 8 weeks.
  Interventions: Behavioral: Sauna Visits

INTERVENTIONS:
Behavioral: Sauna Visits — Weekly 2-hour visits to a sauna in San Francisco by themselves or with one person of their choice for 8 weeks.

SUMMARY:
This pilot trial will test an intervention (sauna visits) targeting reductions in loneliness in adults aged 19-22 years.

Participants will:

* Visit a sauna in San Francisco once per week for 2 hours by themselves or with a friend, for 8 weeks total
* Complete online surveys throughout their participation

The main question this pilot trial aims to answer are:

* To what extent do participants find the study design acceptable?
* To what extent do participants complete the weekly sauna visits?
* To what extent do participants complete the weekly online surveys?

DETAILED DESCRIPTION:
In the U.S. today, emerging adults (i.e., ages 19 to 22) report high levels of loneliness and social isolation, which are significant risk factors for myriad poor health outcomes. This formative period of emerging adulthood is arguably among the most critical of times: it is when the people who comprise our next generation of leaders have some of their earliest opportunities to build their identities as curious about, accepting of, and open to differences from their peers.

Traditional sauna bathing is a social, mental, and physical health practice associated with greater mental wellness and active social engagement. Recent studies also suggest that thermal therapies, including sauna, may reduce depressive symptoms, which contribute to loneliness and social isolation. Sauna bathing is deeply integrated into the social fabric of several cultures, most notably Finland where it serves as a communal activity that fosters social connection and may help reduce loneliness.

ELIGIBILITY:
Inclusion Criteria:

* Aged 19-22
* English-speaking
* Able to provide written informed consent
* Graduated from high school or high school equivalent
* Elevated level of loneliness
* Able and willing to receive study text messages
* Able to attend weekly in-person sauna visits in San Francisco, CA

Exclusion Criteria:

* Self-reported heat intolerance
* Pregnancy, active lactation, or intention to become pregnant during the study period
* Regular use of any nicotine products, including cigarettes, vapes, chewing tobacco, or other forms of nicotine (if use is not regular, must be willing to refrain for 24 hours before and 24 hours after sauna visits)
* Current social heat practices 2 or more times per month (e.g., visiting sauna or hot tub facilities with others present)
* Unwilling to refrain from using marijuana products and alcohol for the 24 hours before and 24 hours after sauna visits
* Unwilling to refrain from heavy exercise on the day of sauna visits
* Any medical condition that, in the opinion of investigators, may increase the risk of sauna use or introduce excessive variance into physiological or behavioral responses to sauna visits
* Use of any medication that might impact thermoregulatory capacity or that, in the opinion of investigators, would increase risk of study participation or introduce excessive variance into physiological or behavioral responses to sauna visits

Ages: 19 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01-03 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Participation Acceptability | 8 weeks
  Average rating on the following net promoter item: "Thinking about everything that participating in this study involved (completing screening activities, visiting the sauna, doing questionnaires), would you recommend participating in this study to a friend or family member looking to reduce their feelings of loneliness?"

SECONDARY OUTCOMES:
Intervention Adherence | 8 weeks
  Proportion of study sauna visits attended (out of 8)
Weekly Survey Completion | 8 weeks
  Proportion of weekly surveys completed (out of 8)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley E Mason, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Osher Center for Integrative Health, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The final IPD dataset will include de-identified self-reported demographic data, self-reported data (e.g., measures of social interaction loneliness), sauna visit completion data, and study assessment completion data.
Time Frame: Beginning 3 months after the publication of results and unending.
URL: https://osf.io/

REFERENCES:
- [Background] Laukkanen JA, Kunutsor SK. The multifaceted benefits of passive heat therapies for extending the healthspan: A comprehensive review with a focus on Finnish sauna. Temperature (Austin). 2024 Feb 25;11(1):27-51. doi: 10.1080/23328940.2023.2300623. eCollection 2024. PMID 38577299
- [Background] Patrick RP, Johnson TL. Sauna use as a lifestyle practice to extend healthspan. Exp Gerontol. 2021 Oct 15;154:111509. doi: 10.1016/j.exger.2021.111509. Epub 2021 Aug 5. PMID 34363927
- See also: Link to online screening survey — http://sealab.ucsf.edu/research